CLINICAL TRIAL: NCT03606096
Title: Randomised, Double-blinded, Open Label Study in Pregnant Women, Exploring the Impact of Acellular Pertussis Vaccination in Pregnancy on the Immunogenicity in Infants Randomized to Receive Either an Acellular (aP) or Whole Cell Pertussis (wP) Vaccine Subsequently
Brief Title: Gambia Pertussis Study (GaPs)
Acronym: GaPs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Oxford (Other); National Institute for Public Health and the Environment (RIVM) (Other Government); Radboud University Medical Center (Other); Imperial College London (Other); University of Turku (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCC 1600
Record Dates: First submitted 2018-07-02; First posted 2018-07-30 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pertussis
Keywords: immune response; impact of acellular pertussis vaccination
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: Eligible pregnant women will be randomized in parallel into one of four groups: two groups will receive maternal Boostrix ® Polio (GSK) the other two groups Tetanus toxoid as per EPI schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the expectant mothers themselves nor members of the clinical trial team assessing the safety or laboratory-based endpoints (immunogenicity and exploratory immunology) will be aware which of these groups the expectant mother has been randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Boostrix IPV - infant acellular Pertussis (TdaP-aP) (Experimental): vaccination of the mother with Boostrix-IPV vaccine which includes the infant acellular pertussis
  Interventions: Biological: Boostrix IPV infant acellular Pertussis
- Boostrix IPV - infant whole Pertussis (Tdap-wP ) (Experimental): vaccination of mother with Boostrix -IPV which includes infant whole cell pertussis
  Interventions: Biological: Boostrix IPV infant whole Pertussis
- TT - infant acellular Pertussis (T-ap ) (Active Comparator): vaccination of mother with TT-which includes infant acellular pertussis
  Interventions: Biological: TT infant acellular Pertussis
- TT - infant whole Pertussis (T-wP) (Active Comparator): vaccination of mother with T which includes infant whole cell pertussis
  Interventions: Biological: TT infant whole Pertussis

INTERVENTIONS:
Biological: Boostrix IPV infant acellular Pertussis — mother is randomized to receive Boostrix ® Polio (GSK) and infant acellular pertussis
  Arms: Boostrix IPV - infant acellular Pertussis (TdaP-aP)
Biological: Boostrix IPV infant whole Pertussis — mother is randomized to receive Boostrix ® Polio (GSK) and infant whole Pertussis
  Arms: Boostrix IPV - infant whole Pertussis (Tdap-wP )
Biological: TT infant acellular Pertussis — mother is randomised to receive Tetanus Toxoid and infant acellular Pertussis
  Arms: TT - infant acellular Pertussis (T-ap )
Biological: TT infant whole Pertussis — mother is randomised to receive Tetanus Toxoid and infant whole Pertussis
  Arms: TT - infant whole Pertussis (T-wP)

SUMMARY:
Currently, there are two types of vaccines available against pertussis (whooping cough), an infectious disease of the respiratory tract that can be extremely serious in very young children.

Both have advantages and disadvantages: The acellular form (aP, mainly used in resource-rich countries) does not appear to offer as long lasting protection, but the whole cell vaccine (wP, mainly used in LMIC) appears to be generally more reactogenic. There is consensus that a "better pertussis vaccine" ought to be designed.

The GaPs trial is part of a series of clinical trials performed by the PERtussIS COrrelates of Protection Europe (PERISCOPE) Consortium, an EU-funded group of investigators which aims to generate knowledge on immune responses to pertussis. A better understanding of human biomarkers of protective immune responses to B. pertussis and its waning immunity is needed to accelerate the design and testing of new pertussis vaccines with a longer duration of protection.

This proposal describes the design and objectives of the clinical trial to be conducted in the Gambia, which is the only site in Africa involved in the consortium and involves the recruitment of 600 mother/infant pairs. Pregnant women will be randomised to receive either the usually recommended tetanus vaccination or a combination vaccine against whooping cough, diptheria, tetanus and polio. Their infants will receive either aP or wP as part of their EPI vaccines, and resulting immune responses will be characterized in detail up to the age of 9 months. The investigators will use immunological assays to investigate the functional humoral and cellular responses to pertussis in infants born to mothers who are randomized to receiving pertussis vaccine in pregnancy or not, and their infants who will receive either aP or wP vaccine.

Our research questions are:

Does vaccination against pertussis in pregnancy have impact on subsequent immune responses to pertussis vaccine and other EPI vaccines in the infants Does vaccination of infants with wP vaccine induce different levels and functionality of antibody and/or T cell responses than vaccination with aP vaccine What is the difference in innate and acquired immunity- as measured with novel systems vaccinology tools- between being vaccinated with wP versus aP?

DETAILED DESCRIPTION:
The investigators are conducting a randomised, controlled, double-blinded, clinical vaccine trial in pregnant women combined with an open-label controlled Phase IV clinical vaccine trial in their infants.

The trial will examine the differences in immunity generated by aP compared with wP in infants at 5 and 9 months of age, and examine the impact of maternal antibodies on the immune response of infants receiving aP or wP vaccines at two, three and four months.

The investigators aim to address two key question: 1. If measures of immunity in infants given aP or wP differ by 5 and 9 months of age; and 2: If and- if so- how maternal pertussis antibodies affect the development and maintenance of immunity to Bordetella pertussis in infants.

Rationale for the trial:

Pertussis (whooping cough) is an infectious disease that can be very serious- particularly in young infants- but preventable through vaccination. There are two types of vaccines: acellular (aP) and whole cell (wP) vaccines, both extensively used worldwide. A clearer understanding of how these two different types of vaccines work is fundamental when considering adjustments or rethinking vaccination strategies and such knowledge will help the future development of new vaccines, given that some LMIC have already introduced aP but the current WHO recommendation still continues to recommend wP vaccine for those who have not yet switched.

Increases in the incidence of pertussis infection, including fatal cases in young infants, have been recently observed in many regions in the world, more likely associated with the use of aP vaccines. As a consequence, it is now recommended in several countries that women should receive aP vaccination in pregnancy so that their high levels of pertussis antibody which will be passed on via the placenta can protect their babies in early life, before the infants have received sufficient doses of pertussis vaccine themselves. However, it is currently unclear if and how maternal antibodies affect long-term immunity to pertussis in infants.

Unlike in the UK, where many women of childbearing age would have received aP vaccine in childhood, in The Gambia, all women would have been primed with wP vaccine as part of the NIP. Hence a study in this group of women is uniquely placed to assess if different priming regimens could have different quantitative and qualitative effects on transplacental antibody transfer for pertussis antibody, providing additional insights in comparison to parallel studies in Europe under the PERISCOPE consortium (PERtussIS COrrelates of Protection Europe).

A better understanding of human biomarkers of protective immune responses to B. pertussis, and its waning immunity is needed to accelerate the design and testing of new pertussis vaccines with a longer duration of protection.

Trial design:

The investigators will recruit 600 mother/infant pairs. Following informed consent, sensitisation and eligibility checks including antenatal ultrasound to date the pregnancy, pregnant women will be randomised to receive either Boostrix IPV (contains antigens against pertussis, tetanus, diphteria and polio)- a vaccine recommended for pregnant women in the UK and other countries where recent pertussis outbreaks have been observed, or the tetanus vaccine routinely recommended for women in LMIC.

Pre vaccination antibody titres will be measured in the women prior to vaccination between 28-34 week gestation and vaccine responses measured subsequently at the time of giving birth. Cord blood will be collected to measure transfer of maternal antibody. Infants will be grouped to receive either aP or wP at 2,3 and 4 months of age, in line with routine EPI programs. Blood samples will be collected from infants prior to vaccination and following doses of vaccines at specific intervals to measure innate and acquired immune responses and followed up until 9 months of age. Infants will be allocated to subgroups for blood tests so that no infant will have between 4 and max 5 episodes of blood sampling up to the age of 9 months.

Samples will be processed for quantitative and qualitative antibody, innate and acquired cellular immune responses. Where available, samples will be stored for further investigations using transcriptomic and epigenetic methodologies. Samples, results and data will be shared with the PERISCOPE consortium members.

ELIGIBILITY:
Inclusion Criteria:

* signed /thumb-printed informed consent for trial participation obtained
* Pregnant women between 18 and 40 years of age inclusive on day of consent
* Singleton pregnancy
* From 28 to 34 weeks gestation inclusive as determined by USS on day of randomization.
* Resident within easy reach of the clinical trial site (no fixed boundaries will be set and such judgements will be made on a case by case basis by members of the field team in discussion with the potential participant, taking into account knowledge of the local transport links and geography)
* Intention to deliver at the health centre related to the Sukuta clinical trial site
* Willingness and capacity to comply with all the study procedures, including those relating to the newborn infant, in the opinion of the principal investigator or delegee.

Exclusion Criteria:

* History of pre-eclampsia or eclampsia
* Gestational diabetes in current pregnancy
* Rhesus negative multigravida
* Grandmultigravida (more than 5 previous pregnancies)
* Previous late stillbirth (defined as loss of pregnancy at any time after 28 weeks gestation)
* Previous low birth weight baby or premature delivery (defined as a delivery before 37 weeks gestation)
* Previous neonatal death (defined as death of an infant within the first 28 days of life)
* Previous delivery of an infant with a known or suspected genetic or chromosomal abnormality
* History of other significant pregnancy related complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected
* History of other significant neonatal complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected
* Smoke cigarettes, alcohol consumption or use of illegal drugs during current pregnancy
* Significant maternal chronic illness including but not limited to hypertension requiring treatment, heart disease, lung disease, neurological disorders including a history of epilepsy or recurrent afebrile seizures, kidney disease, liver disease, anaemia and other haematological disorders (including sickle cell), endocrine disorders including known diabetes mellitus, autoimmunity
* Severe anaemia (less than 7.0g/dL)
* Known Human Immunodeficiency Virus (HIV) or hepatitis B (HBV) virus positive or found to be HIV or HBV positive during screening
* Positive result for syphilis infection on laboratory testing
* Receipt of any vaccine during the current pregnancy or plans to receive any non-study vaccines during the current pregnancy (tetanus toxoid vaccination is not an exclusion and vaccines given during national campaigns if applicable will not generally be exclusions)
* Any other condition judged to significantly increase the risks to either the mother or the infant within the current pregnancy (including relevant history from previous pregnancies)
* History of anaphylactic or severe allergic reactions to previous vaccines or history of anaphylactic or severe allergic reactions in previous offspring (if applicable)
* Receipt of any blood product including human immunoglobulins at any stage during the current pregnancy or plan to receive any blood products during the period or trial participation (receipt or blood products in an emergency or for obstetric reasons will not represent a protocol deviation given such situations are unplanned)
* Receipt of immunosuppressive or immuno-modulatory medication at any stage during the current pregnancy or plan to receive any such medication during the period or trial participation
* Clinically suspected or confirmed congenital or acquired clotting or bleeding disorders or the current receipt of medications known to alter clotting or bleeding
* Current malaria infection (on the day of randomization and vaccination)
* Any clinically significant signs or symptoms of acute illness, significant abnormalities in vital signs, an axillary temperature of greater than 38.0°C or any recorded fever (greater than 38.0°C) in the preceding 24 hours.
* Two or more symptoms (nausea/vomiting, diarrhoea, headaches, fatigue and myalgia) rated as grade 2 and clinically significant on the maternal systemic reactogenicity scale (2 Table 5) present at baseline on the day of vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized
* involuntarily
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will randomize 600 pregnant women at between 28-34 weeks gestation
Enrollment: 600 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-05-18 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
PT specific antibody GMC | 20 weeks
  PT-specific antibody GMC at 20 weeks in infants vaccinated with aP versus wP
PT specific antibody GMC | 9 months
  PT-specific antibody GMC at 9 months in infants vaccinated with aP versus wP

SECONDARY OUTCOMES:
PT specific antibody | at 20 weeks and 9 months
  PT-specific antibody GMC at 20 weeks and 9 months in infants vaccinated with aP versus wP following maternal vaccination with Boostrix ® Polio (GSK) or Tetanus Toxoid.
change in PT, FHA, and PRN antibody concentrations | at 8 and 20 weeks and at 9 months of age
  Proportion with a 2-fold reduction in PT, FHA, and PRN antibody concentrations (measured in cord blood) from baseline at 8, 20 weeks and 9 months of age in aP versus wP primed infants following maternal immunisation with Boostrix ® Polio (GSK) or Tetanus Toxoid
Pertussis antigen-specific memory B-cell | at 8, 16 weeks and at 9 months of age
  Pertussis antigen-specific memory B-cell frequencies at 8,16 weeks and 9 months of age measured by ELISpot in the aP versus wP group following maternal immunisation with aP or Boostrix ® Polio (GSK) or Tetanus Toxoid
Pertussis antigen-specific Th1, Th2 and Th17 responses | at 16 weeks of age of the infant
  Pertussis antigen-specific Th1, Th2 and Th17 responses determined by flow-cytometry and cytokine analysis following antigen-specific culture (the 'Rapid T-cell assay').
PT, FHA and PRN-specific antibody GMC and GMR | at baseline (cord blood baseline) and at 8, 20 weeks and at 9 months
  PT, FHA and PRN-specific antibody GMC and GMR prior to immunisation (cord blood baseline) and at 8, 20 weeks and 9 months of age.
Hib, diphtheria, tetanus, pneumococcal and polio-specific antibody | at 8, 20 weeks and 9 months
  Hib, diphtheria, tetanus, pneumococcal and polio-specific antibody concentrations
Serious adverse events (SAE) in expectant mothers | at 28-34 weeks gestation up to eight weeks from the end of pregnancy.
  Serious adverse events (SAE) in expectant mothers from enrollment at 28-34 weeks gestation up to eight weeks from the end of pregnancy.
local and systemic reactogenicity | within first 3 days of aP administration
  Proportion of mothers 28-34 weeks gestation with local and systemic reactogenicity within the first three days of aP administration
PT specific antibody | at 9 months post delivery
  PT-specific antibody GMC 9 months post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Beate Kampmann, MD, PhD, Principal Investigator — MRC Unit at LSHTM
Locations (1):
- Sukuta Health Centre, Sukuta, City of Banjul, The Gambia

REFERENCES:
- [Derived] Saso A, Froberg J, Jobe H, Eleveld M, Okoye M, Kanteh E, Arns A, van Opzeeland F, Kumado M, Faal A, Roberts E, Fofana ML, Baldeh AK, Conteh K, van Cranenbroek B, Roetynck S, de Jonge M, de Silva TI, Huynen M, Kampmann B, Diavatopoulos DA; GaPs Study Team. Mucosal immune responses to Bordetella pertussis in Gambian infants after maternal and primary vaccination: an immunological substudy of a single-centre, randomised, controlled, double-blind, phase 4 trial. Lancet Microbe. 2026 Jan;7(1):101219. doi: 10.1016/j.lanmic.2025.101219. Epub 2026 Jan 7. PMID 41519134
- [Derived] Saso A, Kanteh E, Jeffries D, Okoye M, Mohammed N, Kumado M, Roetynck S, Jobe H, Faal A, Roberts E, Gageldonk P, Buisman AM, Froberg J, Cavell B, Lesne E, Barkoff AM, He Q, Tanha K, Bibi S, Kelly D, Diavatopoulos D, Kampmann B; Gambian Pertussis Study Team; members of the PERISCOPE consortium. The effect of pertussis vaccination in pregnancy on the immunogenicity of acellular or whole-cell pertussis vaccination in Gambian infants (GaPS): a single-centre, randomised, controlled, double-blind, phase 4 trial. Lancet Infect Dis. 2025 Aug;25(8):909-924. doi: 10.1016/S1473-3099(25)00072-6. Epub 2025 Mar 25. PMID 40154521
- [Derived] Saso A, Kampmann B. What Is the Impact of Maternal Pertussis Immunization in Pregnancy on the Quantity, Quality and Longevity of Infant Vaccine Responses?: A Review of the Current Evidence. Pediatr Infect Dis J. 2025 Feb 1;44(2S):S49-S55. doi: 10.1097/INF.0000000000004692. Epub 2025 Feb 14. PMID 39951075